CLINICAL TRIAL: NCT01320735
Title: Prospective, Multi-Center, Observational Program to Assess Routine Use of Intermittent Adjuvant Deprivation Therapy With Lucrin Depot in Patients With Advanced Prostate Cancer in the Russian Federation
Brief Title: Observational Program to Assess Use of Intermittent Adjuvant Deprivation Therapy With Leuprorelin (Lucrin Depot) in Patients With Advanced Prostate Cancer (PCa) in Russia
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Almedis (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-763
Record Dates: First submitted 2011-02-14; First posted 2011-03-22 (Estimated); Results first posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-06

CONDITIONS: Prostate Cancer
Keywords: Lucrin Depot; intermittent adjuvant regimen; advanced prostate cancer; Leuprorelin
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Advanced PCa: Participants with advanced PCa

SUMMARY:
The objective of this study was to describe treatment patterns of leuprorelin over 2 years using an intermittent, adjuvant regimen in participants with advanced prostate cancer (PCa)

DETAILED DESCRIPTION:
Participants started hormone treatment with Leuprorelin 3.75 mg once every 28 days, subcutaneously (SC) or intramuscularly (IM). Duration of induction therapy was at least 6 months (6-9 months) during which PSA and testosterone levels were measured every 3 months. When PSA decreased by greater than 90% from baseline (PSA less than 10 ng/ml) or became lower than 4.0 ng/ml (for 2 consecutive measurements made at least 2 weeks apart) the participants were included into intermittent hormone therapy regimen group (IAD). Participants with PSA decrease not achieved greater than 90% or less than or equal to 4.0 ng/ml were given either continuous hormone therapy (CAD) or chemotherapy.

Therapy was stopped if participants had PSA decrease greater than 90% from baseline or values less than 4.0 ng/ml after 6-9 months of continuous hormone therapy. PSA and testosterone were measured every 4 weeks. If PSA became greater than or equal to 10.0 ng/ml, hormone therapy was resumed until PSA was less than 4.0 ng/ml for 2 consecutive measurements made at least 2 weeks apart. Duration of hormonal therapy cycle was at least 3 months. Then intermittent treatment was performed according to a similar scheme. PSA and testosterone levels were determined every 12 weeks when hormone therapy was administered and every 4 weeks after it was stopped. The treatment was carried out for 2 years or until Hormone Refractory Prostate Cancer (HRPC) developed.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed advanced PCa meeting the following criteria:

   1. Any Tumor, Node 1, Metastasis 0
   2. Any Tumor, Node 0, Metastasis 1 [according to Tumor Node Metastasis classification 2009]
2. Participants planned for administration of leuprorelin
3. World Health Organization status 0-1
4. Life expectancy at least 2 years

Exclusion Criteria:

1. Contraindications to administration of leuprorelin:

   1. Hypersensitivity to Leuprorelin similar products of protein origin or any of the excipients in drug product composition
   2. Surgical castration
2. Hormone-refractory PCa
3. Presence of another malignant tumor (except skin cancer)
4. Previous administration of hormone therapy with gonadotropin-releasing hormone agonists or antiandrogens
5. Previous administration of radiotherapy or chemotherapy course within 1 month
6. Testosterone level less than or equal to 50 ng/dl (less than or equal to 1.7 mmol/l) at time of inclusion
7. Extremely high level of PSA (greater than or equal to 1000 ng/ml)
8. Other severe diseases in stage of decompensation
9. Other contraindications, that make the participant's participation impossible (by investigator judgment)
10. Previous enrollment in the present program

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with advanced PCa
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Strugovshchikov, MD, Study Director — AbbVie

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: From 300 participants enrolled in the study, data of 17 participants from one of the sites were excluded from analysis because of the impossibility to contact the investigator for data clarification. Hence 283 participants were included in the analysis.
Groups:
- Advanced Prostate Cancer (PCa): Participants with advanced PCa
Period: Overall Study
Arm/Group | Advanced Prostate Cancer (PCa)
Started | 300
Completed | 194
Not Completed | 106
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 13
Not completed — Administrative Reason | 6
Not completed — Progression/Hormone-Refractory Pca | 55
Not completed — Protocol Violation | 1
Not completed — Other | 1
Not completed — No Decrease of Prostate Specific Antigen | 7
Not completed — Investigator Unable to be Contacted | 17

BASELINE CHARACTERISTICS:
Population: Data are of measurements collected from the safety analysis set, defined as all participants who signed an informed consent form and were administered at least one dose of Leuprorelin.
Arm/Group | Advanced PCa
Number analyzed (Participants) | 283
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.4 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 283

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Duration of IAD Regimen Induction Phase
Description: Time period between first injection of leuprorelin and stopping of treatment due to appropriate decrease of PSA as defined in the protocol. The data are reported as mean months +/- standard deviation.
Time Frame: At least 6-9 months after Baseline (enrollment)
Population: Data are of measurements collected from participants who started IAD.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Advanced PCa
Number analyzed (Participants) | 240
Months
  All participants (N=240) | 7.70 (1.25)
  Participants with no progression (N=207) | 7.75 (1.13)
  Participants with progression (N=33) | 7.32 (1.79)

2. Primary Outcome: Mean Duration of Leuprorelin Exposure
Description: Total duration of leuprorelin Intermittent Androgen Deprivation (IAD) regimen was calculated as (Last dose date of Leuprorelin minus first dose date plus 1)/30.4. If the stop date of leuprorelin administration was missing then the date of last attended visit was used. Total duration may include gaps between the cycles. The data are reported as mean months +/- standard deviation.
Time Frame: 24 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Advanced PCa
Number analyzed (Participants) | 283
Months
  All participants | 19.74 (6.39)
  Participants with no progression (N=227) | 21.25 (5.31)
  Participants with progression (N=56) | 13.62 (6.79)

3. Primary Outcome: Mean Duration of Each Leuprorelin Cycle
Description: Duration of each cycle of leuprorelin IAD regimen was calculated as (Date of last dose of cycle of leuprorelin minus start date of cycle plus 1)/30.4. The data are reported as mean months +/- standard deviation.
Time Frame: 24 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Advanced PCa
Number analyzed (Participants) | 283
Months
  All Participants: Cycle 1 (N=282) | 7.63 (1.73)
  All Participants: Cycle 2 (N=238) | 5.60 (2.21)
  All Participants: Cycle 3 (N=61) | 4.64 (1.63)
  All Participants: Cycle 4 (N=7) | 3.44 (1.09)
  All Participants: Cycle 5 (N=1) | 3.30 (NA) — Not applicable as only 1 participant was assessed.
  Participants with No Progression: Cycle 1 (N=226) | 7.68 (1.49)
  Participants with No Progression: Cycle 2 (206) | 5.70 (2.08)
  Participants with No Progression: Cycle 3 (N=52) | 4.72 (1.55)
  Participants with No Progression: Cycle 4 (N=7) | 3.44 (1.09)
  Participants with No Progression: Cycle 5 (N=1) | 3.30 (NA) — Not applicable as only 1 participant was assessed.
  Participants with Progression: Cycle 1 (N=56) | 7.43 (2.49)
  Participants with Progression: Cycle 2 (N=32) | 4.96 (2.84)
  Participants with Progression: Cycle 3 (N=9) | 4.19 (2.08)

4. Secondary Outcome: Number of Participants Who Progressed to Hormone Refractory Prostate Cancer (HRPC)
Description: Progression to HRPC was defined as castrate serum testosterone less than 50 ng/dL or 1.7 nmol/L plus either; biochemical progression (three consecutive rises in prostate specific antigen (PSA) levels one week apart resulting in two 50 % increases over the nadir, with PSA greater than 2 ng/ml) or radiological progression (the appearance of two or more new bone lesions on bone scan or enlargement of a soft tissue lesion using Response Evaluation Criteria in Solid Tumors (RECIST). Data are reported as number of participants with HRPC.
Time Frame: Baseline (enrollment), after 1 year, after 2 years, and 30 days from 2 year visit
Population: Data are of measurements collected from the full analysis set, defined as all participants who received at least one dose of leuprorelin, signed informed consent, did not violate any inclusion/exclusion criteria and attended at least one post-baseline visit.
Measure: Number; unit: Participants
Arm/Group | Advanced PCa
Number analyzed (Participants) | 255
Participants
  All Participants | 36
  Participants who started IAD | 28
  Participants who did not start IAD | 8

5. Primary Outcome: Median Number of Leuprorelin Cycles
Description: The Participants were on IAD regimen and the data are reported as number of cycles with full range.
Time Frame: 24 months
Population: Data are of measurements collected from the safety analysis set, defined as all participants who signed an informed consent form and were administered at least one dose of leuprorelin. However, one participant started continuous hormone therapy and was not included in the analysis.
Measure: Median (Full Range); unit: Cycles
Arm/Group | Advanced PCa
Number analyzed (Participants) | 282
Cycles | 2 [1 to 5]

6. Secondary Outcome: Median Time to Progression of HRPC
Description: Time to progression of HRPC was calculated as date of progression minus date of first dose of leuprorelin. The data are reported as median (full range).
Time Frame: Baseline (enrollment), after 1 year, after 2 years, and 30 days from 2 year visit
Population: as for outcome 4
Measure: Median (Full Range); unit: Months
Arm/Group | Advanced PCa
Number analyzed (Participants) | 255
Months
  All Participants (N=36) | 17.12 [3.00 to 24.80]
  Participants who started IAD (N=28) | 19.10 [5.00 to 24.80]
  Participants who did not start IAD (N=8) | 8.11 [3.00 to 15.40]

7. Secondary Outcome: Median Time to Progression of HRPC in Participants Not Started on IAD Regimen
Description: Time to progression of HRPC was calculated as date of progression minus date of first dose of leuprorelin. A Kaplan-Meier estimate of median time to progression to HRPC and 25% and 75% quartiles along with the 95% confidence interval for median were assessed.
Time Frame: Baseline (enrollment), after 1 year, after 2 years, and 30 days from 2 year visit
Population: Data are of measurements of participants who did not start on IAD regimen.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Advanced PCa
Number analyzed (Participants) | 20
Months | 12.8 [12.8 to 15.4]

8. Secondary Outcome: Median Survival Time
Description: Time to survival was estimated as time from start of leuprorelin up to study completion/discontinuation from the study or date of death. The data are reported as median months with full range.
Time Frame: Baseline (enrollment), after 1 year, after 2 years, and 30 days from 2 year visit
Population: Participants who died while on study were used for analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | Advanced PCa
Number analyzed (Participants) | 4
Months
  All Participants (N=4) | 18.94 [11.80 to 24.80]
  Participants who started IAD (N=2) | 24.44 [24.10 to 24.80]
  Participants who did not start IAD (N=2) | 12.76 [11.80 to 13.80]

9. Other Pre Specified Outcome: Number of Participants Who Received IAD Regimen During the Study
Description: The data are reported as number of participants.
Time Frame: 24 months
Population: Data are of measurements collected from participants who started IAD.
Measure: Number; unit: Participants
Arm/Group | Advanced PCa
Number analyzed (Participants) | 243
Participants
  All participants | 243
  Participants with no progression | 210
  Participants with progression | 33

10. Other Pre Specified Outcome: Number of Participants Who Continued to Take Leuprorelin in IAD Regimen by the End of the Study
Description: The data are reported as number of participants.
Time Frame: 24 months
Population: Data are of measurements collected from participants who started IAD.
Measure: Number; unit: Participants
Arm/Group | Advanced PCa
Number analyzed (Participants) | 243
Participants
  All participants | 69
  Participants with no progression (N=210) | 68
  Participants with progression (N=33) | 1

11. Primary Outcome: Percentage of Participants Who Discontinued From Leuprorelin Administration of IAD Regimen
Description: The data are reported as percentage of participants.
Time Frame: 24 months
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Advanced PCa
Number analyzed (Participants) | 283
Percentage of participants
  Overall Study | 31.4
  Cycle 1 | 15.2
  Cycle 2 (N=240) | 14.6
  Cycle 3 (N=119) | 62.2
  Cycle 4 (N=17) | 64.7
  Cycle 5 (N=1) | 0.0

12. Secondary Outcome: Mean Duration of Treatment-off Time in IAD Regimen
Description: Duration of each leuprorelin free period was calculated as (Date of first dose of leuprorelin [cycle N+1] minus last dose date [cycle N] minus 1)/30.4. If date of last dose of leuprorelin was before the date of study completion/discontinuation then the last leuprorelin free period was calculated as (Date of discontinuation/study completion minus last leuprorelin dose date)/30.4. The data are reported as mean months +/- standard deviation.
Time Frame: Baseline (enrollment), after 1 year, after 2 years, and 30 days from 2 year visit
Population: Data are of measurements collected from participants who started IAD.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Advanced PCa
Number analyzed (Participants) | 243
Months | 7.12 (2.61)

13. Primary Outcome: Number of Participants Who Switched to IAD Regimen by Visit
Description: The data are reported as number of participants.
Time Frame: 24 months
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Advanced PCa
Number analyzed (Participants) | 283
Participants
  Visit 2 After One Year (N=257) | 237
  Visit 3 After Two Years (N=225) | 197

14. Secondary Outcome: Median Percentage of Time Off-treatment During 2 Years IAD Regimen
Description: The total duration of leuprorelin free period was calculated as the sum of all leuprorelin free periods. The data are reported as median percentage of time off-treatment with full range.
Time Frame: Baseline (enrollment), after 1 year, after 2 years, and 30 days from 2 year visit
Population: Data are of measurements collected from participants who started IAD.
Measure: Median (Full Range); unit: Percentage of time off-treatment
Arm/Group | Advanced PCa
Number analyzed (Participants) | 243
Percentage of time off-treatment | 33.45 [0.00 to 67.60]

ADVERSE EVENTS:
Time Frame: From signing of informed consent up to 24 months of observation of treatment period and 30 days of follow up period
Arm/Group | Advanced PCa
Serious Adverse Events (participants affected / at risk) | 13/283
Other Adverse Events (participants affected / at risk) | 73/283
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Advanced PCa (N=283)
DISEASE PROGRESSION (General disorders) | 7
CARDIAC DISORDER (Cardiac disorders) | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1
URINARY RETENTION (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Advanced PCa (N=283)
NASOPHARYNGITIS (Infections and infestations) | 31
BRONCHITIS (Infections and infestations) | 16
PNEUMONIA (Infections and infestations) | 1
DISEASE PROGRESSION (General disorders) | 13
FATIGUE (General disorders) | 5
ASTHENIA (General disorders) | 1
OEDEMA (General disorders) | 1
HOT FLUSH (Vascular disorders) | 12
HYPERTENSION (Vascular disorders) | 2
GYNAECOMASTIA (Reproductive system and breast disorders) | 6
BREAST ENLARGEMENT (Reproductive system and breast disorders) | 4
ACQUIRED HYDROCELE (Reproductive system and breast disorders) | 1
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 1
GASTRITIS (Gastrointestinal disorders) | 3
PEPTIC ULCER (Gastrointestinal disorders) | 2
GASTRIC ULCER (Gastrointestinal disorders) | 1
DERMATITIS (Skin and subcutaneous tissue disorders) | 5
DIABETES MELLITUS (Metabolism and nutrition disorders) | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 3
CARDIAC DISORDER (Cardiac disorders) | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 1
DEPRESSION (Psychiatric disorders) | 1
URINARY RETENTION (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.